CLINICAL TRIAL: NCT05707689
Title: The Impact of Gaming on Functioning Among People With Schizophrenia: a Randomised Controlled Trial (GAME-A)
Brief Title: The Impact of Gaming on Functioning Among People With Schizophrenia
Acronym: GAME-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Collaborators: City of Helsinki (Other)
Responsible Party: Principal Investigator, Maritta Välimäki, Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNITurku
Record Dates: First submitted 2023-01-09; First posted 2023-02-01 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Psychotic Disorder
Keywords: psychotic disorder; gaming; functioning
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A controlled clinical trial with a pragmatic, multi-center, two-arms parallel-group design.
Who Masked: Investigator
Masking Description: Statisticians will be masked. Gaming facilitators, research assistant who collect the data or staff working in the study sites are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gaming (Experimental): Gaming intervention with entertainment video games will be run in small groups (6-10 players) closely monitored by trained gaming facilitators. Pre-scheduled gaming sessions, about 60 minutes each, will be run twice a week over 10 weeks (totally 20 hours).
  Interventions: Behavioral: Entertainment gaming
- Treatment as usual (TAU) (No Intervention): Participants will join usual practices as planned in community services. No specific activities will be organized to them by the research team.

INTERVENTIONS:
Behavioral: Entertainment gaming — If needed, gaming schedule will be tailored based on the participants' individual needs (working, studying, family issues) as long as the total gaming hours will be achieved. Participants are encouraged not to play video games during the study period. Participants' gaming interventions will be monitored carefully and recorded after each gaming session in specific gaming diary.
  Arms: Gaming

SUMMARY:
The goal of this clinical trial is to test whether gaming intervention works well for persons with psychotic disorder. The main question to be answered is whether gaming works well in improving functioning, some other clinical outcomes or causing any adverse effects. Researchers will compare gaming group to usual care.

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate the effectiveness of gaming to improve functioning and clinical outcomes in people with psychotic disorders. Feasibility of the intervention will also be assessed. Our hypothesis are as follows:

Primary hypothesis:

1. Gaming is more effective on improving functioning 3- and/or 6-months follow-ups comparing to usual practices (TAU).

   Secondary hypotheses:
2. Gaming is more effective on improving clinical outcomes and treatment acceptance (symptoms, self-efficacy, the quality of life, drop-out from intervention) at 3-and/or 6-months comparing to usual practices (TAU).
3. Gaming do not cause more adverse effects up to 6 months, especially aggression at 3-and/or 6-months follow-ups comparing to usual practices (TAU).

The effectiveness of the gaming will be assessed using a controlled clinical trial with a pragmatic, multi-center, two-arms parallel-group design. Feasibility will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Finnish speaking
* A formal diagnosis of psychotic disorders (F20-F29, ICD-10; to be identified in medical records or other reliable sources by staff)
* Age between 18 and 60 years old
* Ability to participate in the study based on their own free will
* Ability to provide written informed consent

Exclusion Criteria:

* Clinical diagnostic criteria for a current major depressive, manic or hypomanic episode or mental retardation (ICD-10)
* Severe visual impairment
* Signs or diagnosis of gaming addiction
* Lack of ability to decide one's own participation (under guardianship)
* Substance abuse (other than nicotine dependence)
* Head injury, hemiplegia, or other neurological disorder
* Electroconvulsive therapy (ECT) in the past six months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 356 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Functioning | Day 0, Month 3, Month 6
  The change in functioning will be assessed with the Personal and Social Performance Scale. The instrument includes four domains: a) socially useful activities, b) personal and social relationships, c) self-care, and d) disturbing and aggressive behavior. Difficulty in each area is rated on a single item using a six-point scale (absent, mild, manifest but not marked, marked, severe, or very severe). A global item will be rated by the nurse, ranging from 1 to 100 in ten-point intervals: lower scores indicate poorer functioning.

SECONDARY OUTCOMES:
Major symptoms of mental health | Day 0, Month 3, Month 6
  The symptoms of mental health will be assessed by the Behavior and Symptom Identification Scale®, which focuses on psychopathology and functioning, The instrument is a brief, patient self-reported measure with 24 items, structured based on six sub-scales (Depression and Functioning, Relationships, Self-Harm, Emotional Liability, Psychosis, Substance Abuse). Mean scores for sub-scales and the total score are calculated: the lower the score, the less frequent symptoms/difficulty.
Depressive symptoms | Day 0, Month 3, Month 6
  The severity of depression will be assessed with the Patient Health Questionnaire-9. The instrument includes nine items. The total score of this self-administered questionnaire is calculated. The range of the score vary between 0 and 27: the higher the score, the severe the depression.
Self-efficacy | Day 0, Month 3, Month 6
  Self-efficacy will be assessed using the General Self-Efficacy Scale ith 10 items. Responses of each items are summed up to create a composite score, which ranges grom 10-40: the higher score represent higher self-efficacy.
The quality of life | Day 0, Month 3, Month 6
  The quality of life will be assessed with the Quality of Life Enjoyment and Satisfaction. It is a self-report measure with 15 items. Each question is rated on a 5 point scale from 1 (very poor) to 5 (very good). The first 14 items are summed to form a total score, which can be reported as either the raw score (a maximum 70 points) or as percentage maximum possible, with higher scores indicating greater enjoyment and satisfaction of life. In addition, there is one item that is scored individually from 1 to 5 to describe overall life satisfaction.
Engagement with the intervention | Through intervention completion, an average 3 months
  Number of participants who have dropped out from the intervention (yes/no, n/%), experimental group only
Engagement with the study (%) | Through study completion, an average 6 months
  Number of participants who have dropped out from the study (yes/no, n/%)
Adverse effect: Relapse, a dosage increased | Through study completion, an average 6 months
  Number of participants with a dosage increase reported by staff (yes/no, n/%)
Adverse effect: Relapse, additional medicines prescribed | Through study completion, an average 6 months
  Number of participants with additional medicines prescription reported by staff (yes/no, n/%)
Adverse effect: Symptoms | Through study completion, an average 6 months
  Number of participants with an exacerbation of psychotic symptoms leading to any change in patient management (yes/no, n/%)
Adverse effect: Admission into psychiatric hospital (yes/no) | Through study completion, an average 6 months
  Number of participants admitted in psychiatric hospital (yes/no, n/%)
Adverse effect: The number of hospitalisations | Through study completion, an average 6 months
  The total number of admissions in psychiatric hospital (N)
Adverse effect: The number of hospital days | Through study completion, an average 6 months
  Total number of hospital days (N)
Adverse effect: Violent incidents | Through study completion, an average 6 months
  Number of participants with any violent incidents necessitating staff involvement (whether victim or accused, targeting to another person or property (yes/no, n/%)
Adverse effect: The number of violent incidents | Through study completion, an average 6 months
  Total number of any violent incidents necessitating staff involvement, whether victim or accused, targeting to another person or property (N)
Adverse effect: Self-harming | Through study completion, an average 6 months
  Number of participants with any self-harming behavior (e.g. suicide, an attempt of suicide) (yes/no, n/%)
Adverse effect: The number of self-harm incidents | Through study completion, an average 6 months
  Total number of any self-harming behavior (e.g. suicide, an attempt of suicide)
Adverse effect: Aggression | Day 0, Month 3, Month 6
  Buss-Perry Aggression Questionnaire-Short Form will assess patient aggression with 12 items and four subareas (anger, physical aggression, hostility, verbal aggression). Items are rated on a 5-point scale ranging from 1 ("extremely uncharacteristic of me") to 5 ("extremely characteristic of me"). The value of each item are calculated to form a total score: a higher score indicate higher aggressive behavior.
Adverse effect: Death | Through study completion, an average 6 months
  Death

OTHER OUTCOMES:
Feasibility of the study: Patient refusal | Through study completion, an average 6 months
  Refusal rate (yes/no, n/%)
Feasibility of the intervention | Month 3
  Feasibility of the intervention will be assessed using Feasibility of Intervention Measure, FIM. It includes four items. Responders are asked to rate one of five options (1= completely disagree, disagree, neither agree nor disagree, agree, completely agree). The sum score will ranges from 4 to 16: the higher the score, the better feasibility.
Fidelity of the intervention: The total number of gaming sessions | Through intervention, an average 3 months
  The total number of gaming sessions participated out of 20 (N/%)
Fidelity of the intervention: The total intervention time | Through intervention, an average 3 months
  Total intervention time in hours out of 20 hours (total hours/20, %)
Acceptability of the intervention | Month 3
  Acceptability of the intervention will be assessed using the Acceptability of Implementation Measure, AIM. It includes four items. Responders are asked to rate one of five options (1= completely disagree, disagree, neither agree nor disagree, agree, completely agree). The sum score will range from 4 to 16: the higher the score, the better acceptability of the intervention.
Appropriateness of the intervention | Month 3
  Appropriateness of the intervention will be assessed with the Implementation Appropriateness Measure, IAM. It includes four items. Responders are asked to rate one of five options (1= completely disagree, disagree, neither agree nor disagree, agree, completely agree). The sum score will ranges from 4 to 16: the higher the score, the more appropriate is the intervention.
Implementation process of the novel intervention (qualitative interviews) | Through the study, an average 6 months
  An organizational analysis will be conducted (Consolidated Framework for Implementation Research,CFIR); interviews with nursing staff of the study organisation will be conducted using five major domains: 1) Intervention characteristics (intervention source, evidence strength and quality, relative advantage etc.), 2) Outer setting (patient needs and resources, peer pressure, external policies and incentives, etc.), 3) Inner setting (structural characteristics, culture, implementation climate, etc.), 4) Characteristics of the individuals involved (knowledge and beliefs about the intervention, self-efficacy, individual stage of change, etc.), and 5) Process of implementation (planning, engaging, executing, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Maritta Välimäki, PhD, Principal Investigator — University of Turku
Locations (1):
- City of Helsinki, Helsinki, South Finland, Finland

IPD SHARING:
Plan to Share IPD: No
According to the Ethical Approval, the data will not be shared to other researchers. A meta-data of the study (a general description) will be openly available to researchers.

REFERENCES:
- [Background] Choi WT, Yu DK, Wong T, Lantta T, Yang M, Valimaki M. Habits and Attitudes of Video Gaming and Information Technology Use in People with Schizophrenia: Cross-Sectional Survey. J Med Internet Res. 2020 Jul 22;22(7):e14865. doi: 10.2196/14865. PMID 32459646
- [Background] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Background] Athanasopoulou C, Valimaki M, Koutra K, Lottyniemi E, Bertsias A, Basta M, Vgontzas AN, Lionis C. Internet use, eHealth literacy and attitudes toward computer/internet among people with schizophrenia spectrum disorders: a cross-sectional study in two distant European regions. BMC Med Inform Decis Mak. 2017 Sep 20;17(1):136. doi: 10.1186/s12911-017-0531-4. PMID 28931385
- [Background] Valimaki M, Kuosmanen L, Hatonen H, Koivunen M, Pitkanen A, Athanasopoulou C, Anttila M. Connectivity to computers and the Internet among patients with schizophrenia spectrum disorders: a cross-sectional study. Neuropsychiatr Dis Treat. 2017 Apr 27;13:1201-1209. doi: 10.2147/NDT.S130818. eCollection 2017. PMID 28490882
- [Derived] Valimaki M, Satamo M, Yang M, Vahlberg T. The impact of gaming on functioning among people with schizophrenia: study protocol for a randomised controlled trial (GAME-A). Trials. 2026 Jan 21. doi: 10.1186/s13063-026-09456-2. Online ahead of print. PMID 41566338

DOCUMENTS (1):
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT05707689/ICF_000.pdf